CLINICAL TRIAL: NCT01759498
Title: The Effects of Hydrogen-rich Formulation for Treatment of Sport-related Soft Tissue Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Sergej M. Ostojic, MD, PhD, Head of Human Performance Laboratory, Center for Health Sciences, Serbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 012-12C/4; RPP-3 (Other Grant/Funding Number: NORP Inc.)
Record Dates: First submitted 2012-12-25; First posted 2013-01-03 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Soft Tissue Injuries
Keywords: Inflammation; Pain intensity; Flexibility; RICE protocol; Swelling
MeSH Terms: conditions — Soft Tissue Injuries; Inflammation; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HYDRO 2 (Experimental): Subjects in the second experimental group will follow the procedures of first experimental group with additional administration of hydrogen-rick packs 6 times per day for 20 minutes throughout the study.
  Interventions: Dietary Supplement: HYDRO 2
- ACTIVE (Active Comparator): During the period of 2 weeks subjects will receive traditional treatment protocol after the soft-tissue injury, consisting of RICE protocol during the first 48 h (e.g. rest, ice packs for 20 minutes every 2 hours, compression with elastic bandage, elevation of the injured area above the level of the heart at all possible times) and sub-acute protocol thereafter (e.g. passive stretching 3 times per day for 90 sec, isometric strength exercise with 3 sets with 15 repetitions, 30 min of pain-free weight-bearing exercise).
  Interventions: Dietary Supplement: ACTIVE
- HYDRO (Experimental): Subjects in the first experimental group will follow the PLA procedures with additional administration of oral hydrogen-rich capsules (4 capsules three times per day) throughout the study.
  Interventions: Dietary Supplement: HYDRO

INTERVENTIONS:
Dietary Supplement: HYDRO
  Arms: HYDRO
Dietary Supplement: ACTIVE
  Arms: ACTIVE
Dietary Supplement: HYDRO 2
  Arms: HYDRO 2

SUMMARY:
Since hydrogen therapy in humans seems to be beneficial for treating inflammation, ischemia-reperfusion injury and oxidative stress, it seems plausible to evaluate the effects of exogenously administered hydrogen as an element of instant management of sport-related soft tissue injuries (e.g. muscle sprain, ligament strain, tendonitis, contusion). The main aim of the present study will be to examine the effects of two-week hydrogen-rich oral and topical administration on the inflammation, recovery and functional abilities in competitive male and female athletes after acute soft-tissue injury. During the season 2012/2013 (from February to June) subjects (36 professional athletes) will be recruited and examined by certified sports medicine specialist in the out-patient clinics of the Center for Health, Exercise and Sport Sciences in the first 24 hours after the sport-related soft tissue injury was sustained. The subjects will be allocated to a double-blind design to three randomly assigned trials. During the period of 2 weeks subjects in the placebo group (PLA) will receive traditional treatment protocol after the soft-tissue injury, consisting of RICE protocol during the first 48 h and sub-acute protocol thereafter. Subjects in the first experimental group will follow the above procedures with additional administration of oral hydrogen-rich capsules (4 capsules three times per day) throughout the study. Subjects in the second experimental group will follow the procedures of first experimental group with additional administration of hydrogen-rick packs 6 times per day for 20 minutes throughout the study. Participants will be evaluated at the beginning of the study (e.g. at the time of the injury report), after 7 and 14 days after baseline testing for: a) serum C-reactive protein, plasma viscosity and interleukin 6 level, b) pain intensity during rest and walking, c) degree of joint swelling, d) passive joint flexibility, and, e) subjective side-effects. The investigators expect that the administration of hydrogen will significantly improve inflammation outcomes (e.g. decrease in serum C-reactive protein) as compared to the placebo, with topical hydrogen administration will additionally improve post-injury recovery outcomes (e.g. pain intensity, degree of swelling). These results could support the hypothesis that hydrogen-rich intervention may be included as an element of immediate treatment for sport-related soft tissue injuries.

ELIGIBILITY:
Inclusion Criteria:

* recent history of acute soft-tissue sports injury
* professional athletes

Exclusion Criteria:

* not ambulatory patients
* clinical findings classed as more severe than grade II

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
change in serum C-reactive protein | every week, up to 2 weeks

SECONDARY OUTCOMES:
change in pain intensity during rest and walking | every week, up to 2 weeks

OTHER OUTCOMES:
change in degree of joint swelling | every week, up to 2 weeks
change in passive joint flexibility | every week, up to 2 weeks
change in plasma viscosity | every week, up to 2 weeks
change in serum interleukin 6 | every week, up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sergej M Ostojic, MD, PhD, Principal Investigator — Center for Health, Exercise and Sport Sciences
Locations (1):
- Center for Health, Exercise and Sport Sciences, Belgrade, Serbia

REFERENCES:
- [Background] Ostojic SM. Serum alkalinization and hydrogen-rich water in healthy men. Mayo Clin Proc. 2012 May;87(5):501-2. doi: 10.1016/j.mayocp.2012.02.008. No abstract available. PMID 22560529
- [Background] Jackson MJ. Free radicals generated by contracting muscle: by-products of metabolism or key regulators of muscle function? Free Radic Biol Med. 2008 Jan 15;44(2):132-41. doi: 10.1016/j.freeradbiomed.2007.06.003. Epub 2007 Jun 13. PMID 18191749
- [Background] Ohno K, Ito M, Ichihara M, Ito M. Molecular hydrogen as an emerging therapeutic medical gas for neurodegenerative and other diseases. Oxid Med Cell Longev. 2012;2012:353152. doi: 10.1155/2012/353152. Epub 2012 Jun 8. PMID 22720117
- [Derived] Ostojic SM, Vukomanovic B, Calleja-Gonzalez J, Hoffman JR. Effectiveness of oral and topical hydrogen for sports-related soft tissue injuries. Postgrad Med. 2014 Sep;126(5):187-95. doi: 10.3810/pgm.2014.09.2813. PMID 25295663